CLINICAL TRIAL: NCT02461043
Title: Adjuvant Chemotherapy With Paclitaxel and Cisplatin in Lymph Node-Positive Thoracic Esophageal Squamous Cell Carcinoma: A Randomized Phase 3 Trial
Brief Title: Adjuvant Chemotherapy With Paclitaxel and Cisplatin in Lymph Node-Positive Adjuvant Chemotherapy in the Treatment of the Lymph Node Positive Thoracic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie He, MD.,PhD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-046
Record Dates: First submitted 2015-05-30; First posted 2015-06-03 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; adjuvant chemotherapy; esophageal surgery; paclitaxel
MeSH Terms: conditions — Esophageal Neoplasms | interventions — TP protocol; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): chemotherapy and radiotherapy
  Interventions: Drug: paclitaxel; cisplatin; Radiation: radiation
- Arm B (Active Comparator): radiotherapy
  Interventions: Radiation: radiation

INTERVENTIONS:
Drug: paclitaxel; cisplatin — The adjuvant chemotherapy regimen consisted of paclitaxel 150mg/m2 intravenously (IV) over 3 hours on day 1, followed by cisplatin 50mg/m2 IV on day 2 every 14 days for 4 to 6 cycles.
  Arms: Arm A
Radiation: radiation — radiation

SUMMARY:
Esophageal cancer is a highly aggressive malignancy with a poor overall outcome.

* Five year survival rate after radical esophagectomy is modest at about 40%.The patients with regional lymph node metastases have worse outcome than those without lymph node metastases.
* No standard postoperative adjuvant chemotherapy has ever been established.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent
* histological proof of thoracic esophageal squamous cell carcinoma with negative proximal and distal margins
* node-positive and pathologic stage M0
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients were enrolled 4 to 10 weeks after surgery
* Adequate organ function was required in 2 weeks of registration and was defined as: serum creatinine within normal institutional limit, and creatinine clearance (CrCl) ≥60ml/minute. Aspartate aminotransferase and bilirubin<2 times of upper normal institutional limits

Exclusion Criteria:

* prior chemotherapy or concurrent radiation therapy before esophagectomy
* R1 or R2 resection
* clinically significant hearing loss or symptomatic peripheral neuropathy during initial examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
3 year relapse free survival | 5 years

SECONDARY OUTCOMES:
3 year overall survival | 5 years

OTHER OUTCOMES:
5 year overall survival | 8 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China